CLINICAL TRIAL: NCT06200324
Title: Clinical Outcomes of the Use of Ready-to-Use Parenteral Nutrition in Very Low Birth Weight Newborns in a Fourth-level Neonatal Intensive Care Unit in Cali, Colombia, March 2017-March 2023
Brief Title: Clinical Outcomes of Ready-to-Use Parenteral Nutrition in Low Birth Weight Newborns in Colombia 2017-2023
Acronym: NUMETA
Status: Completed | Type: Observational
Sponsor: Fundacion Clinica Valle del Lili (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Adriana Ballesteros, Neonatologist, Fundacion Clinica Valle del Lili
Other Study IDs: 2023.189
Record Dates: First submitted 2023-11-14; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Very Low Birth Weight Infant
Keywords: parenteral nutrition; premature infants; hydroelectrolytic disorders; plasma glucose concentration; anthropometric measurements
MeSH Terms: conditions — Hyperphagia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ready-to-Use Parenteral Nutrition: Numeta G13E
  Interventions: Other: Ready-to-Use Parenteral Nutrition
- Individualized parenteral nutrition: Individualized parenteral nutrition

INTERVENTIONS:
Other: Ready-to-Use Parenteral Nutrition — In newborns weighing less than 1000 grams, parenteral nutrition is initiated at volumes of 70-80 ml/kg/day up to a maximum volume of 128 ml/kg/day, with a provision of 4 grams/kg/day of protein and a metabolic rate of 12 mg/kg/minute.
  For newborns weighing between 1001-1500 grams, parenteral nutrition is initiated at volumes of 70-80 ml/kg/day up to a maximum of 110 ml/kg/day.
  When enteral intake exceeds 70 ml/kg/day, a gradual decrease in the volume of parenteral nutrition is initiated. We discontinue parenteral nutrition in newborns weighing less than 1000 grams with enteral volume of 120 ml/kg/day, and for those between 1000 grams and 1500 grams, enteral nutrition volume of 100 ml/kg/day.
  Other Names: Numeta G13E
  Groups: Ready-to-Use Parenteral Nutrition

SUMMARY:
The proposed study aims to assess the clinical outcomes of using ready-to-use parenteral nutrition, specifically Numeta G13E, compared to individualized parenteral nutrition in neonates with very low birth weight. Conducted in a level 4 neonatal intensive care unit from March 2017 to March 2023, the study focuses on growth parameters (weight, head circumference, height), growth velocity, and the incidence of complications. The retrospective open-cohort observational design involves a sample of 284 infants, 142 in each group, considering a 95% confidence level and 80% power. The study addresses the need for a local evaluation of the efficacy of ready-to-use parenteral nutrition in this vulnerable population.

DETAILED DESCRIPTION:
Introduction:

Parenteral nutrition enhances nutrition in very low birth weight newborns (<1500 g) who, due to gastrointestinal immaturity, experience delays in obtaining adequate nutrients enterally. Parenteral nutrition (PN) promotes better growth in all anthropometric variables in this population.

However, complications associated with its use have been documented. A commercial method developed to reduce these complications is ready-to-use parenteral nutrition, a three-chamber bag providing a complete mix of nutrients, offering immediate access, quicker initiation of nutrition, and prescription homogenization. These factors aim to achieve better metabolic stability, improved nutritional intake, and weight, height, and head circumference gain.

This study aims to evaluate outcomes with the initiation of ready-to-use parenteral nutrition.

Theoretical Framework:

Advances in favorable clinical outcomes for preterm newborns result from multiple interventions such as cardiorespiratory support and early infection identification. Despite these efforts, morbidity and mortality outcomes remain stagnant. Optimizing nutritional coverage, especially in preterm infants, is one of the objectives to improve outcomes.

Premature infants, due to their immaturity and typically critical clinical condition, require early initiation of parenteral nutrition to guarantee their nutritional needs and reduce the possibility of extrauterine growth restriction. There is also an association between early protein and energy intake and improved neurodevelopment.

While the benefits of early parenteral nutrition initiation in preterm infants are evident, it is classified as a high-risk medication due to potential errors in preparation, leading to biochemical alterations and infection risk. Standardized ready-to-use nutrition is considered a safe alternative, particularly in institutions with limited technological resources.

Commercial preparations like Numeta 13% meet the requirements recommended by the European Society for Pediatric Gastroenterology, Hepatology, and Nutrition (ESPGHAN) for very low birth weight neonates (<1500 g) and extremely low birth weight preterm infants (<1000 g), presenting a cost-effective alternative to individualized preparations.

Despite the proven need for early parenteral nutrition in critically ill neonates, studies reveal variations in protocol adherence, with a significant percentage of units initiating late protein intake and low energy content. Institutional protocols and software utilization could address these challenges.

Continued controversy exists regarding the optimal composition of parenteral nutrition. While individualized nutrition allows adjustments, especially in preterm infants prone to electrolyte imbalances and metabolic control issues, ready-to-use preparations, though less tailored, show no significant differences in complications.

A proposed cohort study aims to assess significant differences between preterm infants receiving individualized and ready-to-use parenteral nutrition locally.

Justification for the Study:

Very low birth weight newborns require multiple supports, including thermal, respiratory, hemodynamic, and nutritional. Ready-to-use parenteral nutrition, with its immediate availability and standardized composition, reduces infection risks.

This study aims to compare clinical outcomes between individualized and ready-to-use parenteral nutrition in terms of metabolic stability, infections, and growth in preterm infants. Existing studies highlight growth delays in preterm infants, associated with poor neurodevelopment and future metabolic and cardiovascular complications. Early trophic stimulation, supported by parenteral nutrition, facilitates a smooth transition with adequate nutrient supply, aiming for appropriate weight gain.

Recognized publications such as ESPGHAN and NICE endorse the use of ready-to-use parenteral nutrition for its safety, immediate availability, and suitability for approximately 85% of patients. Only the remaining 15% may require individual adjustments for specific metabolic issues. An analytical study as proposed would allow local insights into clinical outcomes in neonates receiving individualized vs. ready-to-use parenteral nutrition.

Research Question:

What are the clinical outcomes of using ready-to-use parenteral nutrition compared to individualized parenteral nutrition in very low birth weight neonates in a level 4 Neonatal Intensive Care Unit during the period March 2017-March 2023?

Research Hypotheses:

Alternative Hypothesis: There are differences in anthropometric measurements and complication incidence between very low birth weight patients receiving individualized parenteral nutrition and Numeta G13E ready-to-use.

Null Hypothesis: There are no differences in anthropometric measurements and complication incidence between very low birth weight patients receiving individualized parenteral nutrition and Numeta G13E ready-to-use.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted to the neonatal intensive care unit between March 2017 and March 2023
* Requirement for Parenteral Nutrition.
* Birth weight less than 1500 grams (very low birth weight).

Exclusion Criteria:

* Patients transferred from another hospital with more than 24 hours of life.
* Incomplete follow-up (until 36 weeks corrected age or discharge).
* Major congenital anomalies.

Max Age: 24 Hours | Sex: All
Age Groups: Child
Study Population: Very low birth weight neonates exposed to individualized or ready-to-use parenteral nutrition in a level 4 neonatal intensive care unit during the period from March 2017 to March 2023.
Sampling Method: Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Weight | 36 weeks corrected gestational age or at the time of discharge of the Neonatal Intensive Care Unit (NICU), whichever came first, assessed through study completion, an average of 1 year.
  Weight in grams
Head circumference | 36 weeks corrected gestational age or at the time of discharge of the Neonatal Intensive Care Unit (NICU), whichever came first, assessed through study completion, an average of 1 year.
  Circumference in centimeters
Length | 36 weeks corrected gestational age or at the time of discharge of the Neonatal Intensive Care Unit (NICU), whichever came first, assessed through study completion, an average of 1 year.
  Length in centimeters
Growth velocity - Height | 36 weeks corrected gestational age or at the time of discharge of the Neonatal Intensive Care Unit (NICU), whichever came first, assessed through study completion, an average of 1 year.
  Length in centimeters gained per unit of time
Growth velocity - Weight | 36 weeks corrected gestational age or at the time of discharge of the Neonatal Intensive Care Unit (NICU), whichever came first, assessed through study completion, an average of 1 year.
  Weight in grams gained per unit of time
Growth velocity - Head circumference | 36 weeks corrected gestational age or at the time of discharge of the Neonatal Intensive Care Unit (NICU), whichever came first, assessed through study completion, an average of 1 year.
  Head Circumference in centimeters gained per unit of time

SECONDARY OUTCOMES:
Number of Participants with Electrolyte disorders | Up to 14 days
  Highest serum levels
Number of Participants with Hyperglycemia | Up to 14 days
  Highest serum glucose level
Number of Participants with Bloodstream infections | 36 weeks corrected gestational age or at the time of discharge of the Neonatal Intensive Care Unit (NICU), whichever came first, assessed through study completion, an average of 1 year.
  Bloodstream infections

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Ballesteros, MD, Principal Investigator — Pediatra Neonatóloga FUNDACION VALLE DEL LILI
Locations (1):
- Fundación Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No
No, due to confidentiality issues.

REFERENCES:
- [Background] Rigo J, Marlowe ML, Bonnot D, Senterre T, Lapillonne A, Kermorvant-Duchemin E, Hascoet JM, Desandes R, Malfilatre G, Pladys P, Beuchee A, Colomb V. Benefits of a new pediatric triple-chamber bag for parenteral nutrition in preterm infants. J Pediatr Gastroenterol Nutr. 2012 Feb;54(2):210-7. doi: 10.1097/MPG.0b013e318232f915. PMID 21866057
- [Background] Sirvent M, Calvo MV, Perez-Pons JC, Rodriguez-Penin I, Marti-Bonmati E, Vazquez A, Romero R, Crespo CL, Tejada P; Grupo de Nutricion Clinica de la SEFH. [Best practices for the safe use of parenteral nutrition multi-chamber bags. Spanish Society of Hospital Pharmacist's Clinical Nutrition Group]. Farm Hosp. 2014 Sep 16;38(5):389-97. doi: 10.7399/fh.2014.38.5.8085. Spanish. PMID 25344132
- [Background] Mena KDR, Espitia OLP, Vergara JAD. Management of Ready-to-Use Parenteral Nutrition in Newborns: Systematic Review. JPEN J Parenter Enteral Nutr. 2018 Sep;42(7):1123-1132. doi: 10.1002/jpen.1165. Epub 2018 Apr 27. PMID 29701872
- [Background] Kreissl A, Repa A, Binder C, Thanhaeuser M, Jilma B, Berger A, Haiden N. Clinical Experience With Numeta in Preterm Infants: Impact on Nutrient Intake and Costs. JPEN J Parenter Enteral Nutr. 2016 May;40(4):536-42. doi: 10.1177/0148607115569733. Epub 2015 Feb 5. PMID 25655621
- [Background] Kriz A, Wright A, Paulsson M, Tomlin S, Simchowitz V, Senterre T, Shepelev J. Cost-Consequences Analysis of Increased Utilization of Triple-Chamber-Bag Parenteral Nutrition in Preterm Neonates in Seven European Countries. Nutrients. 2020 Aug 20;12(9):2531. doi: 10.3390/nu12092531. PMID 32825528
- [Result] Wittwer A, Hascoet JM. Impact of introducing a standardized nutrition protocol on very premature infants' growth and morbidity. PLoS One. 2020 May 21;15(5):e0232659. doi: 10.1371/journal.pone.0232659. eCollection 2020. PMID 32437423
- [Result] Brennan AM, Kiely ME, Fenton S, Murphy BP. Standardized Parenteral Nutrition for the Transition Phase in Preterm Infants: A Bag That Fits. Nutrients. 2018 Feb 2;10(2):170. doi: 10.3390/nu10020170. PMID 29393903
- [Result] Riskin A, Shiff Y, Shamir R. Parenteral nutrition in neonatology--to standardize or individualize? Isr Med Assoc J. 2006 Sep;8(9):641-5. PMID 17058418
- [Result] Smolkin T, Diab G, Shohat I, Jubran H, Blazer S, Rozen GS, Makhoul IR. Standardized versus individualized parenteral nutrition in very low birth weight infants: a comparative study. Neonatology. 2010;98(2):170-8. doi: 10.1159/000282174. Epub 2010 Mar 16. PMID 20234142
- [Result] Díaz Cuesta, E., & Celis Castañeda, L. A. (2022). Prevalencia de la restricción de crecimiento extrauterino y factores de riesgo asociados en recién nacidos con peso menor de 1500 gramos en una unidad de cuidado intensivo neonatal de Bogotá (Colombia). Universitas Medica, 63(2). https://doi.org/10.11144/Javeriana.umed63-2.prce
- [Result] Osegueda-Mayen JR, Sarmiento-Aguilar A. Standarized parenteral nutrition in the NICU: Case Report and composition analysis of the three chamber bag. Acta Pediatr Mex. 2022;43(3):167-73.
- [Result] Setia MS. Methodology Series Module 1: Cohort Studies. Indian J Dermatol. 2016 Jan-Feb;61(1):21-5. doi: 10.4103/0019-5154.174011. PMID 26955090